CLINICAL TRIAL: NCT05353686
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Trial Investigating the Effect of 4 Weeks Bi-daily Dosing of XEN-D0501 on Blood Glucose Reduction as add-on to Metformin in Patients With Diabetes
Brief Title: A Trial Investigating the Effect of 4 Weeks Dosing of XEN-D0501 on Blood Glucose Reduction in Patients With Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pila Pharma (Industry)
Collaborators: Biomapas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PP-CT02; 2018-001880-22 (EudraCT Number)
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Efficacy; Safety; Pharmacokinetics; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a 4 weeks randomised, double-blind, placebo-controlled, parallel-group, prospective trial. Each subject will be randomised to 1 out of 2 possible treatment arms and treated for four weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treatment is blinded for subjects, care provider and investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive an oral tablet containing no active drug twice daily
  Interventions: Drug: Placebo
- XEN-D0501 (Active Comparator): Subjects in the XEN-D050 arm will receive an oral tablet containing 4 mg/tablet of IMP, twice daily
  Interventions: Drug: XEN-D0501

INTERVENTIONS:
Drug: Placebo — Subjects in the placebo arm will receive an oral tablet containing no active drug twice daily
  Arms: Placebo
Drug: XEN-D0501 — Subjects in the XEN-D0501 arm will receive an oral tablet containing 4 mg/tablet of IMP twice daily
  Arms: XEN-D0501

SUMMARY:
This is a randomised, double-blind, placebo-controlled, parallel-group trial investigating the effect of 4 weeks bi-daily dosing of XEN-D0501 on blood glucose reduction as add-on to metformin in patients with diabetes mellitus type 2 where life style changes and treatment with metformin has failed to effectively reduce blood glucose concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must give his/her signed and dated informed consent before any trial-related activities. Trial-related activities are any procedures that would not have been performed during the normal management of the subject
2. Diagnosis of type 2 diabetes mellitus
3. In treatment with a stable metformin dose during the last three months, but no other anti-diabetic drugs
4. HbA1C (glycosylated haemoglobin A1C): 6.5-10 %
5. Age above 25

Exclusion Criteria:

1. A subject with a history of significant multiple drug allergies or with a known or suspected allergy to the trial product or any medicine chemically related to the trial product, as judged by the Investigator.
2. A subject who has a clinically significant abnormal ECG at screening, as judged by the investigator.
3. A subject who has participated in any other trials involving investigational products within the 3 months preceding the start of dosing.
4. A subject who has donated any blood or plasma in the past month or in excess of 500 mL within 1 month preceding screening.
5. A subject who has a significant history of alcoholism or drug/chemical abuse as per investigator's judgement.
6. A subject with mental incapacity or language barriers which preclude adequate understanding or cooperation, who is unwilling to participate in the trial, or who in the opinion of their general practitioner or the Investigator should not participate in the trial.
7. Surgery or trauma with significant blood loss within the last 2 months prior to dosing.
8. A subject with a clinically significant abnormal haematology or biochemistry tests at screening visit, as judged by the Investigator considering the underlying disease.
9. Current treatment with drugs known to interfere with glucose metabolism such as systemic corticoids and monoamine oxidase inhibitors (MAO) inhibitors.
10. Haemoglobin < 6.2 mmol/l (<99.8 g/l), total leukocyte count < 3.0 x 109/l, thrombocytes <100 x 109/l, serum creatinine levels ≥ 126 μmol/l (male) or ≥ 111 μmol/l (female), bilirubin > 3 x ULN, alanine aminotransferase > 2 x the upper limit of normal (ULN), alkaline phosphatase > 2 x ULN, one re-test within a week is permitted.
11. Previous participation (randomisation) in this trial.
12. Any condition that would interfere with trial participation or evaluation of results, as judged by the investigator and/or sponsor
13. Recurrent major hypoglycaemia or hypoglycaemic unawareness, as judged by the Investigator.
14. Females of childbearing potential (i. e. not post-menopausal ≥ 12 months or surgically sterilised) who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral hormonal contraceptives (p-pills), implantants, transdermal patches, p-ring or depot injection, sexual abstinence or vasectomised partner). A male subject who is sexually active and has not been surgically sterilised must be informed that he must ensure that his partner practices effective contraception, as stated above, or he must refrain from sexual intercourse during the trial and until 90 days after completion of the trial. This is to prevent the possibility of a pregnancy from spermatocytes that can potentially be damaged by trial medication.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | 4 weeks of treatment
  Fasting blood glucose after four weeks of bi-daily dosing of XEN-D0501

CONTACTS AND LOCATIONS:
Overall Officials: Dorte X Gram, PhD, Study Director — Pila Pharma
Locations (10):
- Lithuania (10):
  - Kristavita, JSC, Jonava
  - "Auki sveikas" ("A klinika"), Kaunas
  - Saules seimos medicinos centras, JSC, Kaunas
  - Kaunas City Polyclinic / Dainava Outpatient Clinic, Kaunas
  - Kedainiai Hospital / Outpatient Department, Kėdainiai
  - A. Navickas Outpatient Clinic, Klaipėda
  - Karoliniskiu Outpatient Clinic, Vilnius
  - Vilnius University Hospital Santaros Clinics / Family Center Department, Vilnius
  - Vilnius University Hospital Santaros Clinics, Vilnius
  - Vaidotas Urbanavicius Sole Proprietary Enterprise, Vilnius

IPD SHARING:
Plan to Share IPD: No